CLINICAL TRIAL: NCT04581798
Title: Attachment Loss Levels, Periodontal Indices, and Sulcus Bleeding Indices in Patients With Obstructive Sleep Apnea: a Cross-sectional Study
Brief Title: Periodontal Disease in Patients With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-2020
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Sleep Apnea of Adult; Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss
Keywords: Obstructive sleep apnea; Periodontal disease; Periodontal attachment loss; Bleeding on probing; Plaque index
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA: Patients with OSA confirmed by polysomnography, aged 35-65
- Non-OSA: Patients without OSA aged 35-65

SUMMARY:
Investigators hypothesize that in patients with obstructive sleep apnea (OSA) the severity of periodontal disease is significantly higher compared to patients without OSA in every aspect, including PI, PD, CAL and BOP. The number of lost teeth is hypothesized to be also higher in patients with obstructive sleep apnea.

Purpose: evaluation of periodontal status in patients with obstructive sleep apnea.

An analytical cross-sectional study will be conducted at the Department of Therapeutic Dentistry of the Sechenov University, Moscow.

Investigators are planning to recruit 100 patients: 1) patients with OSA confirmed by polysomnography -75 participants aged between 35 and 65; 2) patients without OSA -25 participants of a similar age.

Patients with obstructive sleep apnea syndrome will be sub-divided into three sub-groups according to OSA severity: 2A group - patients with mild apnea severity; 2B group - patients with medium apnea severity; 2C group - patients with severe apnea.

All participants will undergo a dental examination including the following parameters: plaque index (PI; Silness & Loe, 1964), bleeding on probing (BOP), and touch depth of the pocket (PD), the level of clinical attachment loss (CAL). Investigators will also evaluate the number of lost teeth.

DETAILED DESCRIPTION:
Periodontal disease is a chronic inflammatory disease which is associated with an increased risk of many diseases, including bone and cardiovascular disease (Adamkiewicz et al., 2018). The high prevalence and severity of periodontal inflammatory diseases is a current problem in dentistry. A growing body of literature suggests that there is a link between periodontitis and systemic diseases. Nevertheless a cause-and-effect relationship has not been established yet for most of the diseases, and the mediators of the association are still being identified (Bui et al., 2019). In recent years, several studies have revealed a possible link between periodontitis and obstructive sleep apnea (OSA). The main oral symptom of OSA is dry mouth due to oral breathing, which is a significant risk factor for periodontal disease. Chronic periodontitis is characterized by the destruction of the supporting tissues of the teeth through complex cascades of inflammatory responses, and OSA seems to share common pathways, acting synergistically (Ryan Price et al., 2020).

The purpose of the study is to evaluate the periodontal health in patients with obstructive sleep apnea (OSA).

Within an analytical cross-sectional study 150 patients will be examined: 75 patients with obstructive sleep apnoea and 25 patients without OSA.

The diagnosis of sleep apnea will be set after the standard polysomnography in the Domino program. The severity of OSA will be determined according to AHI index.

Patients with obstructive sleep apnea syndrome will be sub-divided into three groups according to sleep apnea severity: 2A group - patients with mild sleep apnea severity; 2B group - patients with medium sleep apnea severity; 3С group - patients with severe sleep apnea.

After confirming the diagnosis of obstructive sleep apnea patients undergo dental examination. Investigators will use a manual periodontal probe to provide basic periodontal examination.

The amount of plaque accumulated in cervical part of the teeth will be registered by the plaque index (PI; Silness & Loe, 1964). The activity of the inflammation will be assessed with use of Bleeding on probing index (BOP). The Pocket Touch Depth (PD) will and the level of clinical attachment loss (CAL) will be recorded. The number of lost teeth will also be estimated.

Potential risk factors for periodontal disease will also be evaluated (body weight index (BMI), smoker status).

ELIGIBILITY:
Inclusion Criteria:

Patients with obstructive sleep apnea

Exclusion Criteria:

Pregnancy and lactation diabetes mellitus coronary heart disease medications associated with xerostomia chronic infectious diseases.

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of the Somnology Center, healthy volunteers recruited from Sechenov University staff.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | baseline
  distance from the cemento-enamel junction (CEJ) to the base of the clinical pocket.
  Measurement takes place with a periodontal probe. Taken together, the probing depth plus the distance from the gingival margin to the CEJ comprises the clinical attachment level

SECONDARY OUTCOMES:
bleeding on probing (BOP index) | baseline
  presence or abscence of bleeding within 10 seconds after probing.
pocket depth (PD) | baseline
  Measure the pocket depth of the groove between your gums and teeth by placing a dental probe beside your tooth beneath your gumline, usually at several sites throughout your mouth.
Silness-Loe plaque index (PI). | baseline
  Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The indices for the following six teeth may be grouped to designate the index for the group of teeth: 16, 12, 24, 36, 32, 44. The index for the patient is obtained by summing the indices for all six teeth and dividing by six.

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No